8-Week Atopic Dermatitis (AD) Treatment Study NCT03386032 April 27, 2018

# **CLINICAL STUDY PROTOCOL**

Title: 8-Week Atopic Dermatitis (AD) Treatment Study

Study Number: CSD2017168

Date Issued: April 27, 2018

Expected Start Date: December 6,2017

Expected Completion Date: July 15, 2018

Test Facility: Wake Research Associates, LLC WR-ClinSearch, LLC

3100 Duraleigh Rd., Suite #304 6035 Shallowford Road, Suite #109

Raleigh, NC 27612 Chattanooga, TN 37421 Phone: 919-781-2514

**Sponsor Facility:** Procter and Gamble Company

11510 Reed Hartman Highway

Cincinnati, OH 45241

### **Sponsor and Investigator Concurrence**

e-mail: rkrause@clinsearch.com

I have reviewed the attached protocol and its associated documents. This clinical study will be conducted in compliance with Federal, state, and local government regulations, guidelines, and standards applicable to such studies including, but not limited to, those relating to ICH E6 and Good Clinical Practices Guidelines, including Informed Consent. The Investigator agrees to abide by the terms of this protocol.

| Sponsor: | | Work Phone: | Alternate Phone: |
|---|---|---|---|
| Debora Whittenbarger, B.S.N., R.N.<br>Clinical Trial Manager<br>e-mail: whittenbarger.dj@pg.com | date | 513-626-1620 | 513-368-4551 |
| Dawn Yeomans, PhD<br>Clinical Scientist<br>e-mail: yeomans.dj@pg.com | date | 513-498-4518 | 315-982-4636 |
| Laurie Moulton, MS<br>Statistician<br>e-mail: moulton.lt@pg.com | date | 513-626-0215 | |
| Suska Bentz, AS<br>Data Manager<br>e-mail: bentz.si@pg.com | date | 513-626-3912 | 513-293-3942 |
| Michael Marmor B.S. Imaging Coordinator e-mail: marmor.mj@pg.com Test Site Investigators | date | 513- 626-0140 | 513-382-3348 |
| rest Site Investigators | | | |
| Adnan Nasir, MD, PhD<br>Principal Investigator, Raleigh Site<br>e-mail: anasir@wakeresearch.com | date | 919-781-2514 | |
| | | 423-698-4584 | |

# **TABLE OF CONTENTS**

| I. | Objective | 2 |
|------|-------------------------------------|-----|
| II. | Background | 3 |
| Α | | |
| В | , 5 | |
| III. | Study Population | |
| C | | |
| VI. | Subject Accountability | 8 |
| Α | | |
| В | • | |
| C | | |
| | ). Illness and Medication Reporting | 8 |
| VIII | . Other Study Documentation | 9 |
| Α | Protocol Amendments | 9 |
| В | Protocol Deviations | 9 |
| C | Study Monitoring | 9 |
| | ). Additional Data | 9 |
| Χ. | Investigator's Responsibilities | 10 |
| Α | Informed Consent / Assent | 10 |
| В | Final Investigator's Report | 10 |
| | ). Record Retention | 11 |
| Е | | |
| F | . IRB Review and Approval | 1 1 |
| XI. | Attachments | 11 |
| Α | . Appendices | 11 |
| В | Data Collection Forms (DCFs) | 12 |
| C | C. Safety Letter | 13 |

# I. Objective

The primary objective of this study is to demonstrate the clinical efficacy of the Sponsor's experimental eczema cream treatment containing formula relative to a basic moisturizer in condition improvement as measured by

SCORAD (scoring of atopic dermatitis). The secondary objective is to demonstrate the clinical efficacy of the Sponsor's experimental eczema cream treatment containing a formula relative to a basic moisturizer in condition improvement as measured by PGA (physician's global assessment), EASI (eczema area and severity index), and individual lesion assessment by the extent and severity components of SCORAD. The tertiary objective is to demonstrate the clinical efficacy of the Sponsor's experimental eczema cream treatment containing formula relative to a basic moisturizer in condition improvement as measured by Qualify of Life (QoL) and self-assessment questionnaires. The quaternary objective is to understand skin health profiles as measured by biomarker analysis from tape strip samples.

# II. Background

Atopic dermatitis (AD) is a chronic inflammatory skin disease characterized by disruption of epidermal barrier function that results in intense pruritus, sleep disturbances, and subacute and chronic eczematous lesions. AD is the most common cause of chronic inflammatory skin disease and is a major cause of morbidity and suffering, affecting up to 30% of children, and increasing in prevalence throughout the world. It is estimated that the direct cost of AD in the US alone may be as high as \$3.8 billion every year.

The current therapy of AD is reactive, where the flares are treated through symptomatic management with topical corticosteroids and calcineurin inhibitors. Given that these medications have long-term side-effects, and given the chronically relapsing immunopathogenic nature of AD, there is an imperative need for safer anti-inflammatory medications. The aim of this study is to provide clinical performance data to support eczema indication claim on package for the PG Ventures medicated skin program.

# A. Study Design

This is an approximately 9-week, 7-visit, randomized, double blind, parallel comparison study consisting of a 7-12 day washout phase followed by an 8-week treatment phase. This study has currently been enrolling for approximately 4 months; full enrollment under the initial IRB approved protocol dated October 26, 2017 has not yet been achieved. The following changes to the initially approved protocol will be implemented as strategies to fully enroll the study as well as to finish the study with a more complete dataset due to a higher number of early subject withdraws than was anticipated in the statistical considerations of sample size. Changes to the study population, inclusion criteria, and enrollment strategy from the initial protocol are as follows:

- Revise inclusion criteria to the following:
  - Omit criteria of VAS, PGA and area coverage (BSA)
  - Revise SCORAD criteria to >=18
  - All other inclusion criteria (antihistamine use, sun exposure, absence of other clinical findings and negative pregnancy test, if applicable) remain the same
- In keeping with the current study design of balancing blacks and non-blacks within each of the 2 test sites, invite back the non-blacks that were previously disqualified, repeat study qualification procedures (Screening + washout), and grade these subjects again at Baseline against the revised inclusion criteria appearing above.

Note: Previously disqualified non-black subjects will be scheduled to visit the test site(s) en mass, meaning all previously disqualified subjects would be seen within the same 1-2 days so that they would be screened and placed on a 7 day washout within the same 1-2 days, and return for their Baseline visit within the same 1-2 days. After all "repeat" subjects have completed their Baseline visit, the Sponsor will review their visual assessment grades (SCORAD, PGA, EASI) and select subjects for randomization into the study using SCORAD criteria >= 18 as minimum entrance criteria, in accordance with the above revised inclusion criteria. Subjects will meet all other inclusion/exclusion criteria as stated in the Protocol. These subjects may remain on washout up to an additional 5 days past the day of their Baseline visit while the Sponsor selects subjects for randomization.

Increase the number of subjects randomized into the study from the initial protocol-specified 62
up to 71 subjects.

**Note:** After review of recruitment observations from this study and data from previous studies, these additional 9 subjects that may be enrolled are to be non-black.

This study will now be conducted among up to **71** male and female subjects aged 12 to 65 years old (inclusive) and executed by one clinical research company utilizing 2 of their test sites as a strategy to fully enroll the study with subjects meeting all revised inclusion/exclusion criteria. Enrollment of black subjects is now capped at the 31 black subjects who have been enrolled. It will be stipulated that there will only be 1 grader of record at each of the 2 test sites who will grade all subjects at each site at every time point.

At Screening and Enrollment, subjects deemed qualified for this phase of the study will be provided with bar soap and body lotion to use for all their skin cleansing and moisturization needs during the washout phase. Subjects will be instructed to refrain from using any other products on their body (excluding the face) including topical corticosteroids, ointments, lotions, sunscreens, etc., must refrain from using shampoo or conditioning products that contain known anti-microbial or anti-inflammatory agents (e.g. anti-dandruff shampoo), and refrain from using any other medications indicated for atopic dermatitis other than the study provided products. Normal facial or hair care products are permitted however they must NOT contain anti-bacterial ingredients (e.g. antidandruff shampoo, acne products, etc.).

At Baseline, start of treatment phase, after visual grading (SCORAD, PGA, EASI) has been completed, the Sponsor will review subjects' visual grading data against the revised, minimum inclusion appearing in this protocol and Protocol Amendment #001. Subjects deemed by the Sponsor qualified (communicated via email from Clinical Trial Manager to Test Site Study Staff) to participate in this study will have one primary lesion and one secondary lesion identified by the Study Dermatologist following the principle that the lesions are from the representative affected areas of the body (preferably the primary from limbs), at the developing phase, not resolution phase, and 2cm or greater. All efforts will be made to identify the primary lesion from limbs (for individual lesion assessment using extent and severity components of SCORAD), and the secondary lesion not having blisters and/or drainage present as determined by the study PI or designee (for both individual lesion assessment using extent and severity components of SCORAD and for tape stripping procedures).

The 4 corners of both the primary and secondary lesions will be marked with "L" brackets using a permanent marker. Subjects will be given a permanent marker and instructed to remark their sites at home each time after bathing or showering for the duration of their study participation. Dermatological lesion assessments and imaging of the primary and secondary lesions will be conducted at Baseline, Weeks 2 4, and 8. Subjects will be randomized and balanced into one of the 3 treatment groups based on severity as defined by their SCORAD grade. Treatment groups and a caption of their application regimens are as follows:

- Desonide will be provided in a tube. Subjects will be instructed to apply this product only to their lesions using the "Finger Tip Method." Subjects will also be given a lotion (same as Vehicle) and instructed to apply the lotion to the remaining unaffected body skin (whole body including face);
- Vehicle and the Sponsor's experimental cream treatment groups will be provided as a tube and lotion (same treatment in both the small treatment tube and the large lotion tube) for blinding purposes. Subject instructions for product application will be the same as for the Desonide group.

**Note:** Five minutes after applying both the lesion treatment and lotion products, if desired, subjects will be allowed to apply their own facial moisturizer and make up over the study treatments.

To help maintain blinding, products will be concealed in an opaque bag. Subjects will be instructed to bring their products with them in the opaque bag to every visit and to refrain from discussing their study participation with other subjects. Subjects will also be asked to complete a daily diary to record their twice daily treatment applications and any medications taken and to bring their diaries with them to every visit.

Study measurements will be conducted at the time points indicated in the table below. Subjects will acclimate with their AD lesion sites exposed to air for at least 30 minutes under office environment conditions prior to any study procedures being performed. Product application and compliance checks as well as dermatologic evaluations (incl. AEs) will be conducted at each subsequent visit following Baseline to ensure the subject's condition does not become extensively worse. For the sake of subject safety, subjects who drop from the study will have the reason(s) for their dropping documented, will be asked to return their study products and diaries to the test site, and as part of their study exit visit procedures be evaluated for SCORAD at the time of their dropping. Additionally, these subjects, will be asked to continue to come to the test site for the remaining study visits for SCORAD evaluations only, if willing, and have AE/Medication changes for the remainder of the study documented.

# B. Study Schedule (listed in procedure order)

| Study<br>Activities | Screen/<br>Enroll,<br>start of<br>washout | Base<br>line | WK<br>1 | WK<br>2 | WK<br>4 | WK<br>6 | WK<br>8 |
|---|---|---|---|---|---|---|---|
| Study Day | -7 to -12 | 1 | 8 | 15<br>3 | 29<br>4 | 43 | 57<br>6 |
| Informed Consent/Assent + Confidentiality Agreement (Appendices IC/Assent + CA) | X | 1 | 2 | 3 | 4 | 5 | 6 |
| Informed Consent for Photo Release-<br>declination does not impact<br>enrollment (Appendix ICPHOTO) | х | | | | | | |
| INCL/EXCL/DEMO<br>(DCF'S INCL, EXCL, DEMO) | X | | | | | | |
| Body system assessment per Test Site SOP's (Appendix SCREENPE) | X | | | | | | |
| Screening labs per Wake SOP's & urine pregnancy test (Appendix SCREENLABS) | x | X | X | X | x | x | X<br>Preg-<br>nancy<br>only |
| Qualify (DCF QUALIFY) | X | | | | | | |
| Distribute bar soap, lotion for washout period (weigh before and after distribution) and Subject Instructions for the washout period (App INWO) | x | | | | | | |
| Acclimate 30-minutes with lesions exposed to air (office environment) prior to all visual assessments | | X | | X | x | | x |
| Pre-visit Compliance Check & Med Hx update/ changes in medications (Appendix QVISITPROCEDURES & DCF CON-MED) | | x | X | X | х | х | х |
| Query subjects for compliance with pre-visit restrictions and instructions | | X | X | X | X | X | X |
| Physician's Global Assessment, whole body (Appendix and DCF PGA) | | X | | X | X | | X |
| SCORAD, Whole Body<br>(Appendix and DCF SCORAD) | | X | | X | x | | Х |
| SCORAD <u>Lesion</u> Evaluation only,<br>extent and severity of primary and<br>secondary lesions<br>(Appendix SCORAD and DCF SCORAD<br>LESION) | | x | | x | х | | х |
| EASI lesion evaluation, whole body (Appendix and DCF EASI) | | X | | X | X | | х |
| Study Activities (DCF Name) (Appendix Name) Sponsor Review of Visual Grading | Screen/<br>Enroll,<br>start of<br>washout | Base<br>line | WK<br>1 | WK<br>2 | WK<br>4 | WK<br>6 | WK<br>8 |
| Data for Study Qualification – selected subjects approved via email to Test Site Staff (EASI, SCORAD, PGA) | | x | | | | | |

| | ī | | T | T | | T |
|---|---|---|---|---|---|---|
| Qualify (DCF QUALIFY_ADD) | X | | | | | |
| Identify and mark/remark primary and | | | | | | |
| secondary lesions | X | Х | X | Χ | Х | Х |
| (app SITEDIAG) | | | | | | |
| Medical History and Habits and | | | | | | |
| Practices Questionnaire | X | | | | | |
| (DCF's H & P and Med Hx) | | | | | | |
| Tolerability Questionnaire | X | х | x | x | x | x |
| (Appendix and DCF Tolerability) | ^ | ^ | ^ | ^ | ^ | ^ |
| Dlqi/Poem/Bother/Qol/Self- | | | | | | |
| Assessment Questionnaires | X | Х | X | X | X | X |
| (Appendices and DCF SAQ 1) | | | | | | |
| Consumer OAR Questionnaires | Х | х | Х | X | Х | х |
| (DCF SAQ2-1, SAQ2-2, SAQ2-3) | | | | | | |
| Digital Image of primary and | X | | Х | Χ | | Х |
| secondary lesions (App Imaging) | | | | | | |
| Tape Stripping, secondary and adjacent non-lesion site (Appendix | Х | | Х | | | x |
| TSSQUAME) | ^ | | ^ | | | ^ |
| Randomize/distribute test products | | | | | | |
| and diaries | X | | | | | |
| 1:1 subject instruction and supervised | | | 1 | 1., | | |
| product application coaching session | X | X | X | Х | Х | |
| Distribute/collect/review diaries | | | | Х | | |
| weigh products, refresh bar soap prn | X | | | Collect | | |
| (Appendices DIARY, DCF CON_SUM) | Distrib<br>Unit #1 | | | Unit #1<br>Lotion | | X |
| _ , | Treatment | Х | X | & | X | Final |
| | and lotion | | | Distrib | | collect |
| | | | | Unit #2<br>Lotion | | |
| 45-minute Consumer Interview, 6-8 | | | | LULIUIT | | |
| willing subjects selected & interviewed | | | | | | |
| by Sponsor rep from 1 test site | | Х | | | | X |
| (Appendix Discussion Guide) | | | | | | |
| | | | | | | t . |

# III. Study Population

A sufficient number of non-black male and female subjects aged 12-65 (inclusive) diagnosed as having AD and otherwise generally healthy will be recruited and/or re-screened if previously disqualified from the general Raleigh, North Carolina and Chattanooga, Tennessee populations in order to fully enroll the study with up to **71** subjects. Enrollment of black subjects is now capped at the 31 black subjects who have been randomized. Subjects will be recruited based on their ability to meet the inclusion/exclusion criteria and their willingness to comply with all study requirements, restrictions and instructions.

Prior to study start all prospective subjects

Will read and sign:

-Informed Consent/Assent if underage, Confidentiality Agreement, and Informed Consent for Photo Release (Appendix IC/ASSENT, CA, and ICPHOTO)

Will be screened for eligibility to participate based on:

- DCF INCL (all answers must be "yes" to qualify)
- DCF EXCL (all answers must be "no" to qualify)
- DEMO
- DCF CON MED
- SCREENLABS
- QUALIFY

At Screening and Enrollment, if a prospective subject is admitted or excluded from the study, this information will be recorded on DCF QUALIFY. Enrolled subjects will be given bar soap, lotion, verbal and written instructions and restrictions to follow during the washout phase (Appendix INTRWO). At Baseline, if a subject is admitted or excluded from the study, this information will be recorded on DCF QUALIFY\_ADD. Qualified subjects at Baseline will be randomized into one of the 3 treatment groups, given verbal and written instructions and restrictions to follow, and daily diaries to complete during the treatment phase (Appendices INTRTRT and DIARY).

# IV. Study Materials

### A. Study Products

The products listed in the table below will be tested during this study. Test products will be stored in a locked room under usual and customary office building conditions. Unit #1 test products (eczema cream and whole body lotion) will be distributed to qualified subjects at Baseline. Subjects will apply their assigned treatments twice daily as directed by their product labels and subject instructions (Appendix INTRTRT).

| Test Product Regimen | Rationale | Observations |
|---|---|---|
| Small tube to apply to lesions twice daily and large lotion tube to apply to whole body except lesion sites – same product both containers | Test product | 34 |
| Small tube to apply to lesions twice daily and large lotion tube to apply to whole body except lesion sites – same product both containers | Control Product | 17 |
| 0.05% Desonide (tube) to apply to lesions twice daily in a small tube and vehicle lotion in a large tube to apply to whole body | Rx control | 11 |

At Weeks 1-6, subjects will be supplied with eczema cream tubes in sequential order (Unit #s 2-6) enough to last until their next study visit. At Week 4, Unit #1 body lotion tube will be collected and subjects will be given Unit #2 body lotion to last for the remaining 4 weeks of the study. All product containers will be weighed pre-distribution and after each collection to assess subjects' consistency of and compliance with product usage.

Supplemental products will be assigned a #5000 series number and will distributed as needed; supplemental product numbers will be assigned using the Sponsor's balance and assignment program.

# B. Product Safety Statement

This study meets the ethical requirements stipulated by the International Conference of Harmonization and Guidelines for Good Clinical Practices for Research Involving Human Subjects. Appropriate safety testing has been completed; risk assessments justify the placement of the test products in this study considering product concentration(s) and frequency of treatment as set forth in the protocol.

# C. Packaging, Labeling, and Shipping of Test Products

The Sponsor will send all test products directly to the clinical facility prior to the start of the study in compliance with current Good Manufacturing Practices. A sample of how the products will be labeled appears in Appendix Label. The quantity of all study material shipped to the clinical facility will be documented on a shipping and receiving form, included within the shipment (DCF SHIP\_REC).

# D. Return of Study Products

Upon completion of the study, the Investigator or his/her designee will assure that all test products (completely used, partially used, or unused) will be returned to the Sponsor at the address listed below. Product accountability will be appropriately documented on DCF SHIP REC.

The Procter & Gamble Company Mason Business Center 8700 S. Mason Montgomery Rd, DV3 5J5 Mason, OH 45040-9462 ATTN: Ryan Nichols Phone: 513-256-1668

# V. Study Procedures

Study procedures will be performed as presented in the following appendices and at the times indicated in the study schedule table listed in Section II.B.

- SCREENPE
- SCREENLABS
- SCORAD
- PGA
- EASI
- SITEDIAG
- DLQI
- POEM
- BOTHER
- IMAGING
- TSSQUAME
- DISCGUIDE

# VI. Subject Accountability

### A. Subject Identification

Subjects will be assigned a permanent 4-digit number (consecutive, beginning with #2001) during the consent process. Subjects will be assigned a permanent consecutive randomization number (beginning with #201) once they have qualified to participate in the treatment phase of the study.

# B. Subject Early Withdrawal

A subject may voluntarily withdraw from the study at any time for any reason. If a subject experiences a problem that they perceive to be related to study participation, or if test facility personnel deem it necessary, the Investigator is responsible to take appropriate action. The Investigator, or designee, will complete a Subject Drop (DCF DROP) form for any subject withdrawal or discontinuation prior to the end of the study. Subjects who withdraw after study initiation will not be replaced.

### C. Adverse Events

Subjects will be evaluated at each visit for Adverse Events using the Common Terminology Criteria for Adverse Events for Skin & Subcutaneous Tissue Disorders (CTCAE) as outlined in the Appendix TOLERABILITY.

The Investigator or designee will complete the DCF AE to record any Adverse Event (AE) that occurs during the study, regardless of relationship to treatment. The Investigator must review and sign the completed form associated with each specific AE.

The Investigator or designee will notify the Clinical Trial Manager within 24 hours of any unexpected and/or serious AE's and notify the IRB within 3 days of any serious adverse events or any events that are related to product treatment or study procedures. The Clinical Trial Manager will notify the Study Toxicologist following the Sponsor's SOP for AE reporting. In the event of multiple adverse events related to test product usage, the Clinical Trial Manager, Clinical Scientist & Study Toxicologist will work with the PI to determine the appropriate course of action up to and including study suspension.

# D. Illness and Medication Reporting

Subjects will be questioned at each visit about their general health and medications as well as their tolerability of the test products (Appendix TOLERABILITY) by a qualified medical professional such as a nurse or physician's assistant. Any adverse changes to their general health will be recorded on DCF AE. Any changes in their medications (prescription or OTC not previously recorded), will be documented as a concomitant medication on the DCF CON\_MED form. Responses to the tolerability questionnaire will be recorded on DCF TOLERABILITY.

# VIII. Other Study Documentation

#### A. Protocol Amendments

If it becomes necessary to modify this protocol, the modification will be documented by a protocol amendment. Amendments will be initiated by the Sponsor and signed by the Investigator or designee and by all the appropriate representatives of the Sponsor who are directly impacted by the change. All amendments will be consecutively numbered, describe any changes being made and the rationale behind the changes. Amendments cannot be implemented until written IRB approval is obtained.

#### B. Protocol Deviations

If a significant deviation from the final protocol occurs, it is the responsibility of the Investigator or designee to notify the Clinical Trial Manager or designee as soon as possible once the deviation is noted and no later than 24 hours after the occurrence. All deviations and subsequent notification will be documented on the Deviation Log (DCF CONDEVERR) for the subject affected. If a deviation affects multiple subjects, it will be recorded on the tab in the eCRF database titled Study Notes.

# C. Study Monitoring

The Investigator will permit a representative of the Sponsor to visit the facility during the course of the study to monitor study progress and to observe all study procedures. During these visits, the Investigator will permit the monitor to inspect all forms and corresponding subjects' records to verify adherence to the protocol. The study monitor will also be permitted to review and verify test materials and any Investigator-generated or Sponsor-generated study documents. The monitor will document and discuss this visit with the Investigator or his designee including any problems that are to be resolved.

#### D. Additional Data

Daily outdoor relative humidity and temperature at the test facility will be recorded during the test period on a site provided data collection form. Acclimation room conditions (temperature controlled office environment conditions) will be recorded at 9 am and 3 pm (+/- 1 hour) each study day at Baseline, Weeks 2, 4, and 8.

# E. Investigator and Site Qualification

After review of the Investigator's CV, the Investigator is qualified to conduct this study based on education, training, and experience conducting similar studies with similar test products and/or methods within the past 2 years. Further, the Investigator remains in good standing with US Governmental agencies regulating the conduct of clinical studies and has agreed via his/her signature on Page 1 of this protocol to conduct this study according to GCP/ICH guidelines. The Investigator has agreed to maintain a list of any personnel to which the Investigator delegates his/her responsibilities and has agreed that selected delegates will have demonstrated they are capable and qualified to perform such functions. A list of all delegates and their responsibilities will be maintained and a copy of this list will be provided to the Sponsor in the Investigator's final report.

The test site has adequate facility space and work processes including current, comprehensive, applicable SOP's, access to sufficient number of prospective subjects meeting the study required demographics, the required equipment and instruments (or Sponsor has agreed to supply), and sufficient qualified staff possessing current and applicable training records, the correct skill sets, any required professional licensure (Study Physician and assisting health professionals as required by state law) to conduct this study in compliance with all Federal, State and local regulations, GCP/ICH guidelines, and according to the protocol. Additionally, the test site has a history of low staff turnover which will increase the likelihood that the quality of study and method conduct will be sustained over the entire in-life portion of the study.

# VII. Data Management and Statistical Analysis

#### A. Data Collection

Data entered directly into the Sponsor's eCRF system will be considered source data. If an independent eCRF database is used (one that is not on the server (i.e., one that is on a dedicated instrument computer for direct data capture)), then data will be backed up nightly to another storage location (i.e., flash drive, CD, external hard drive, etc.). This can be done either by using the "export all" function under the reports tab and placing the files on a location not on the computer or by copying the database to a location not on the computer (i.e., flash drive, CD, external hard drive, etc.). Instrumentation that has a separate data collection system (i.e., not eCRF) needs data backed up daily following the directions in the corresponding instrument appendix, and this data system will be considered source data.

If the eCRF is not available, all study data will be written directly on the paper CRF as source data and recorded into the eCRF when it is available. It is the responsibility of the Investigator or designee to ensure that all source documents and data collection forms are completed, maintained according to Good Clinical Practices, and retained in the study records. This includes assuring that all study documents are filled in completely, entered into the eCRF system and 100% Quality Control reviewed for accuracy in transcription.

All grading direct data entry errors in the eCRF system will be corrected where possible. When the correction is not possible within the eCRF system the error will be documented in the eCRF ComDevErr form. Included in this error documentation should be the error that occurred and the resolution. Errors to be documented are improperly entered subject numbers, invalid grades or instrument data and failure of equipment calibration. It is the responsibility of the Study Investigator or a designee to review the data error record to ensure errors are captured correctly and are easily understood.

### B. Data Transfer

Following study completion and prior to submission of the Clinical Study Summary, the test facility will give sponsor-requested electronic data files, legible copies of the documents (i.e., DCF's) not entered into electronic format to the Data Manager. Original source documents reside with the study facility.

# C. Statistical Analysis

The Statistical Analysis plan for this study is detailed in Appendix STATS.

# X. Investigator's Responsibilities

### A. Informed Consent / Assent

Prior to study participation, all subjects will be informed as to the type of study, the procedures to be followed, the general nature of the products being tested, and any known or anticipated adverse reactions that might result from participation. Each subject must read, comprehend, and sign the informed consent (Appendix IC) before participating in this study. The informed consent will contain all of the basic elements of outlined in ICH E6. For subjects considered to be "underage" following each test site's state laws, study staff will obtain written documentation of parental permission and written documentation of child's willingness to participate through written assent (Appendix ASSENT).

# B. Final Investigator's Report

The Investigator or designee will submit a study report to the Sponsor within 4 weeks following study completion or termination. This report should include:

- Investigator's designee of authority statement and signature for specific tasks, e.g., designation by investigator to a qualified staff person to enroll subjects.
- Personnel list of responsibilities (including any non-Test Site Facility personnel)
- Copy of original Monitor Signature Log and Delegation Signature Log
- Records of the study site visits by the Sponsor
- Documentation that the Investigator has reviewed and approved all subject data for the study
- Documentation by Investigator that all subjects were provided a copy of the Informed Consent

- Number of subjects screened for eligibility
- Number of subjects entering and completing the study
- Number of subjects that withdrew from the study and reasons for withdrawal
- Any deviations or changes/amendments to the protocol
- Summary of adverse events
- Clinical judgments relative to any significant adverse events and their disposition; any alterations in treatment due to adverse events
- Notes to file
- Data transfer
- Forms disposition
- Documentation that source documents transcribed to eCRF have been verified
- Signed and dated quality assurance statement ensuring protocol compliance

### D. Record Retention

The Investigator or designees will retain all study records for a minimum of 5 years. After a minimum of 5 years, the test facility will notify the Sponsor before destroying retained study records.

# E. Confidentiality

All information (photographs, medical information and data evaluations, etc.) concerning the subject that is obtained in connection with this study will be kept confidential. The sponsoring company, governmental regulatory agencies and the Institutional Review Board (IRB) will have access to the study records: however, they will be coded to protect the subject's confidentiality.

# F. IRB Review and Approval

The study will not begin prior to the receipt of written confirmation of approval by the IRB and any relevant regulatory authority. It is the responsibility of the Investigator to obtain the IRB approval (per the U.S. Code of Federal Regulations, Title 21, Part 56 and applicable ICH guidelines) for the protocol, amendments, informed consent, subject information sheet, questionnaires, and advertising materials used to recruit study subjects, if appropriate. A copy of the IRB approval letter along with a list of the IRB members who acted on this protocol and a statement that the IRB is in compliance with current ICH E6 and Good Clinical Practices (GCP) guidelines will be provided to the Clinical Trial Manager.

It is the Investigator's responsibility to promptly report to the IRB all changes to the research activity and all unanticipated problems involving the risk to human subjects.

#### XI. Attachments

#### A. Appendices

| IC/ASSENT | Informed Consent/Assent for Minors |
|---|---|
| ІСРНОТО | Informed Consent for Photo Release |
| CA | Confidentiality Agreement |
| FITZSKIN | Fitzpatrick Skin Type |
| SCREENPE | Body System Assessment (Wake SOP's) |
| CONSENSUS | Outline of Consensus Grading Activities |
| SCREENLABS | Screening Labs Blood Draw and Urine Pregnancy Test Procedure |
| INTRWO | Subject Instructions for the Washout Phase |
| QVISITPROCEDURES | Procedures to be Conducted at Every Visit |
| SCORAD | Severity Scoring of Atopic Dermatitis |
| EASI | Eczema Area and Severity Index |
| PGA | Physician's Global Assessment |
| SITEDIAG | Identify and Mark Lesions & Non-Lesion |

| INTRTRT | Subject Study Instructions for Treatment Phase |
|---|---|
| DIARY | Daily Product Application Diary |
| TOLERABILITY | Instructions for Completion of Tolerability Questionnaire |
| DLQI | Description and Instructions for Completion of Dermatology Life Quality Index |
| POEM | Description and Instructions for Completion of Patient Oriented Eczema Measure |
| BOTHER | Description and Instructions for Completion of Bother Measure |
| IMAGING | Instructions for Obtaining Digital Image of Designated Lesion |
| TSSQUAME | Tape Strip Sampling Procedure |
| DISCGUIDE | Consumer Interview Discussion Guide |
| STATS | Statistical Analysis Plan |
| LABEL | Sample Product Labels |

# B. Data Collection Forms (DCFs)

| INCL | Inclusion Criteria |
|---|---|
| EXCL | Exclusion Criteria |
| DEMO | Demographics |
| CON_MED | Concomitant Medications |
| QUALIFY | Qualification at Enrollment |
| PGA | Physician's Global Assessment |
| SCORAD | Severity Scoring of Atopic Dermatitis |
| SCORADLESION | Objective Severity Scoring of Primary & Secondary Atopic Dermatitis Lesions |
| EASI | Eczema Area and Severity Index |
| QUALIFY_ADD | Qualification at Baseline |
| MEDHX | Medical History |
| HAB_PRAC | Habits & Practices |
| SAQ-1 | DLQI / POEM / Bother Questionnaires |
| SAQ-2-1, 2-2, 2-3 | Consumer Self-Assessment Questionnaire – (OAR) |

| TOLERABILITY | Tolerability Questionnaire |
|--------------|----------------------------------|
| COMDEVERR | Comment, Deviation and Error Log |
| CON_SUM | Product Consumption |
| DROP | Subject Drop Form |
| AE | Adverse Event Form |
| SHIP_REC | Ship and Receiving Log |

# C. Safety Letter

To be provided by the Sponsor.